CLINICAL TRIAL: NCT01747278
Title: The Safety and Effectiveness of Trimethoprim/Sulfamethoxazole as Pneumocystis Carinii Pneumonia (PCP) Prophylaxis in Patients With Connective Tissue Diseases
Brief Title: Study of Trimethoprim/Sulfamethoxazole as PCP Prophylaxis in CTD Patients
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Fengchun Zhang, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-CTD-PCP
Record Dates: First submitted 2012-12-09; First posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-12

CONDITIONS: Pneumonia, Pneumocystis; Prevention & Control
Keywords: Pneumocystis carinii pneumonia; prophylaxis; trimethoprim/sulfamethoxazole
MeSH Terms: conditions — Pneumonia, Pneumocystis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (No Intervention): Patients were not treated with Trimethoprim/Sulfamethoxazole (TMP/SMX).
- TMP/SMX (Experimental): Patients received Trimethoprim/Sulfamethoxazole (TMP/SMX) 80 mg/400 mg p.o. every day as PCP Prophylaxis.
  Interventions: Drug: Trimethoprim/Sulfamethoxazole

INTERVENTIONS:
Drug: Trimethoprim/Sulfamethoxazole — Oral Trimethoprim/Sulfamethoxazole 80 mg/400mg once daily for 12 weeks.
  Other Names: Septra
  Arms: TMP/SMX

SUMMARY:
Evaluation the efficacy and safety profile of trimethoprim/sulfamethoxazole as Pneumocystis carinii pneumonia (PCP) prophylaxis in Patients With Connective Tissue Diseases (CTD) treated with high-dose glucocorticoids and immunosuppressive agents.

Open-labeled, randomized, prospective single-center clinical trial. Observation period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years with informed consent
* SLE, Sjögren syndrome, Polymyositis or Dermatomyositis, defined by consensus classification criteria
* concomitant high dose glucocorticoid, defined as >1mg/kg/d prednisone or equivalent
* concomitant cyclophosphamide, cyclosporine or mycophenolate mofetil

Exclusion Criteria:

* Pregnant or lactating
* WBC< 4×10^9/L，PLT<100×10^9/L
* Serum ALT or AST > 2 times upper limit of normal
* Serum creatinine > 1.5 mg/dL
* Severe hepatic, hematological, gastrointestinal, pulmonary, cardiovascular, neurological, endocrine or cerebral disease
* Active infection, including HIV, HCV, HBV, tuberculosis or PCP
* concomitant antibiotics other than trimethoprim/sulfamethoxazole
* Patient with malignancy
* Drug allergy, especially trimethoprim/sulfamethoxazole

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-06 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Documented PCP infection | 12 weeks.
  Documented Pneumocystis carinii pneumonia infection: defined as documentation of Pneumocystis from a properly obtained specimen (induced sputum, bronchoalveolar lavage, or biopsy) in a patient with clinical manifestations compatible with PCP.

SECONDARY OUTCOMES:
PCP-related mortality | 12 weeks
  PCP-related mortality at the end of week 12.
All cause mortality | 12 weeks
  All cause mortality at the end of week 12.
Other infections | 12 weeks
  Infections other than PCP throughout the study period.
PCP-related hospitalization | 12 weeks
  PCP-related hospitalization throughout the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Fengchun Zhang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Deptment of Rheumatology, Peking Union Medical College Hospital, Beijing, China